CLINICAL TRIAL: NCT06838572
Title: Effect of Remote Local Peripheral Nerve Cooling on Pain of Arterial Puncture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HH123
Record Dates: First submitted 2025-02-09; First posted 2025-02-20 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-02

CONDITIONS: Acute Pain
Keywords: Skin cooling; arterial puncture; analgesia
MeSH Terms: conditions — Acute Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, patient-assessor blinded
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Skin cooling to 20°C (Experimental): The superficial skin of the right brachial plexus (superficial skin of the axillary artery at the junction of the right pectoralis major and biceps) cooled to 20°C for 15 minutes.
  After cooling, 1ml 2% lidocaine was injected into the superficial skin of the right radial artery.
  After local anesthesia, right radial artery puncture catheterization was performed.
  Immediately after the puncture, warm air at 35°C was applied to the cooling treatment area for 10 minutes, and the target temperature was the surface temperature of the area before cooling treatment.
  Interventions: Procedure: Skin cooling to 20°C
- Skin cooling to 15°C (Experimental): The superficial skin of the right brachial plexus (superficial skin of the axillary artery at the junction of the right pectoralis major and biceps) cooled to 15°C for 15 minutes.
  After cooling, 1ml 2% lidocaine was injected into the superficial skin of the right radial artery.
  After local anesthesia, right radial artery puncture catheterization was performed.
  Immediately after the puncture, warm air at 35°C was applied to the cooling treatment area for 10 minutes, and the target temperature was the surface temperature of the area before cooling treatment.
  Interventions: Procedure: Skin cooling to 15°C
- Skin cooling to 8°C (Experimental): The superficial skin of the right brachial plexus (superficial skin of the axillary artery at the junction of the right pectoralis major and biceps) cooled to 8°C for 15 minutes.
  After cooling, 1ml 2% lidocaine was injected into the superficial skin of the right radial artery.
  After local anesthesia, right radial artery puncture catheterization was performed.
  Immediately after the puncture, warm air at 35°C was applied to the cooling treatment area for 10 minutes, and the target temperature was the surface temperature of the area before cooling treatment.
  Interventions: Procedure: Skin cooling to 8°C
- No skin cooling (Placebo Comparator): The superficial skin of the right brachial plexus does not need to be cooled. After waiting 15 minutes, 1ml2% lidocaine was injected into the superficial skin of the right radial artery.
  After local anesthesia, right radial artery puncture catheterization was performed.
  There is no need to warm the radial artery after catheterization.
  Interventions: Procedure: No skin cooling

INTERVENTIONS:
Procedure: Skin cooling to 20°C — According to the group, copper parts at a constant temperature of 20°C were placed on the superficial skin of the brachial plexus for 15 minutes.
  Arms: Skin cooling to 20°C
Procedure: Skin cooling to 15°C — According to the group, copper parts at a constant temperature of 15°C were placed on the superficial skin of the brachial plexus for 15 minutes.
  Arms: Skin cooling to 15°C
Procedure: Skin cooling to 8°C — According to the group, copper parts at a constant temperature of 8°C were placed on the superficial skin of the brachial plexus for 15 minutes.
  Arms: Skin cooling to 8°C
Procedure: No skin cooling — According to the group, copper parts at room temperature (23°C) were placed on the superficial skin of the brachial plexus for 15 minutes.
  Arms: No skin cooling

SUMMARY:
In this project, volunteers will be recruited to cool the superficial skin of the axillary brachial plexus away from the puncture point, resulting in local peripheral nerve cooling, and observe its impact on the pain of arterial puncture.To explore the local peripheral nerve cooling treatment can produce controllable and reversible analgesic effect even if away from the wound, and provide a new nonpharmaceutical analgesic mode for clinical.

DETAILED DESCRIPTION:
Arterial puncture is a common cause of iatrogenic pain and anxiety, which can lead to stress and arterial spasm, leading to puncture failure.Clinicians usually use pharmacology to treat acute pain, but it is often accompanied by circulatory and respiratory depression, abnormal coagulation function, edema, pruritus, nausea, vomiting, constipation, addiction, etc., which can lead to death, and doctors strictly restrict the use of indications.In addition to drugs, electrical, light, mechanical or thermal stimulation can produce local reversible blocking effect of the peripheral nerve.Temperature is a simple, controllable and reversible physical factor.Current studies have shown that cooling the peripheral nerve to 10-15°C for 10 minutes can relieve pain, and numbness can occur after 15 minutes.These results suggest that cooling the peripheral nerve of sensory innervation in the remote trauma area can reduce nerve conduction velocity and signal amplitude, and provide a new method for non-pharmaceutical analgesia.Local peripheral nerve cooling therapy is an attractive approach to blocking nociceptive information because it is non-addictive, reversible, and allows simultaneous electrophysiological monitoring of the blocked nerve.In this project, volunteers will be recruited to cool the superficial skin of the axillary brachial plexus away from the puncture point, resulting in local peripheral nerve cooling, and observe its impact on the pain of arterial puncture.To explore the local peripheral nerve cooling treatment can produce controllable and reversible analgesic effect even if away from pain stimulation, and provide a new nonpharmaceutical analgesic mode for clinical.

ELIGIBILITY:
Inclusion Criteria:

1. 18 ~ 65 years old;
2. ASA I-II level;
3. Patients with perioperative invasive arterial blood pressure monitoring;
4. Right-handed;
5. Allen test was normal (palm color quickly turned red or returned to normal within 10 seconds after release of ulnar artery pressure);
6. Participate voluntarily and be able to understand and sign informed consent.

Exclusion Criteria:

1. Patients with a history of musculoskeletal, vascular, neurological or psychiatric disorders;
2. Patients with a history of diabetes or other systemic diseases
3. Patients who used any analgesic medication within the month before and during the study;
4. Patients with a history of smoking, alcohol or drug addiction;
5. Paraesthesia, scar, redness, damage, rash, etc. exist in the skin of the patient in the test area;
6. Patients whose surgical area overlaps with the cooling treatment or puncture area;
7. Female subjects are menstruating.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Pain Scale (VAS) score of arterial puncture procedure | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  The larger values of the Visual Analogue Pain Scale (VAS) score of local anesthetic injection and the Visual Analogue Pain Scale (VAS) score of arterial puncture catheterization were taken as the Visual Analogue Pain Scale (VAS) score of the process of arterial puncture catheterization.(VAS ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable)

SECONDARY OUTCOMES:
Pressure pain threshold | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  Before the start of cooling therapy, 5 minutes into cooling therapy, 15 minutes after the start of cooling therapy, and 10 minutes after rewarming, the handheld algometer is used to measure the Pressure Pain Threshold (PPT) at the following locations:
  The midpoint of the ulna and radius at the wrist joint of both forearms (as bony pressure pain points) The brachioradialis muscle on the lateral side of the forearm (as muscular pressure pain points) Unit: Kilograms-force per square centimeter (kg/cm²)
Pressure pain tolerance | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  Before the start of cooling therapy, 5 minutes into cooling therapy, 15 minutes after the start of cooling therapy, and 10 minutes after rewarming, the handheld algometer is used to measure the Pressure Pain Tolerance (PTO) at the aforementioned locations.
  Unit: Kilograms-force per square centimeter (kg/cm²)
The average perfusion | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  Before the administration of local anesthesia, during the process of local anesthesia, after the completion of local anesthesia, before arterial puncture, during the arterial puncture procedure, and after the completion of arterial puncture, the patient is instructed to maintain a calm state and lie in a supine position with the left arm abducted. Under these conditions, the Region of Interest (ROI) is outlined using laser speckle technology, and the average perfusion of this area is measured.
The median perfusion | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  Before the administration of local anesthesia, during the process of local anesthesia, after the completion of local anesthesia, before arterial puncture, during the arterial puncture procedure, and after the completion of arterial puncture, the patient is required to remain calm and in a supine position with the left arm abducted. Under these conditions, the Region of Interest (ROI) is outlined using laser speckle technology, and the median perfusion of this area is measured.
The maximum perfusion | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  Before the administration of local anesthesia, during the process of local anesthesia, after the completion of local anesthesia, before arterial puncture, during the arterial puncture procedure, and after the completion of arterial puncture, the patient is required to remain calm and in a supine position with the left arm abducted. Under these conditions, the Region of Interest (ROI) is delineated using laser speckle technology, and the maximum perfusion of this area is measured.
The minimum perfusion | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  Before the administration of local anesthesia, during the process of local anesthesia, after the completion of local anesthesia, before arterial puncture, during the arterial puncture procedure, and after the completion of arterial puncture, the patient is required to remain calm and in a supine position with the left arm abducted. Under these conditions, the Region of Interest (ROI) is delineated using laser speckle technology, and the minimum perfusion of this area is measured.
The approximate depth of the right brachial plexus. | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  Perform ultrasound localization of the right axillary artery depth before the start of hypothermia treatment.
  Unit: millimeters (mm).
Depth of the Right Radial Artery | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  Place the ultrasound probe at a position 1 cm proximal to the right radial styloid process to measure the distance from the skin surface to the center of the right radial artery at the following time points:before the start of cooling, 5 minutes into cooling, 15 minutes after the start of cooling, and 10 minutes after rewarming.
  Unit: Millimeters (mm)
Peak Systolic Velocity (PS) | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  The maximum blood flow velocity in the right radial artery during the systolic phase of the cardiac cycle is measured at the following time points: before the start of cooling, 5 minutes into cooling, 15 minutes after the start of cooling, and 10 minutes after rewarming. The ultrasound probe is placed 1 centimeter proximal to the styloid process of the right radius, reflecting the artery's ability to transport blood.
  Unit: Centimeters per second (cm/s)
End Diastolic Velocity (ED) | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  The blood flow velocity at the end of the diastolic phase in the right radial artery is measured at the following time points: before the start of cooling, 5 minutes into cooling, 15 minutes after the start of cooling, and 10 minutes after rewarming. The ultrasound probe is placed 1 centimeter proximal to the styloid process of the right radius, to assess changes in blood flow.
  Unit: Centimeters per second (cm/s)
Time-Averaged Maximum Velocity (TAMAX) | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  The highest average blood flow velocity in the right radial artery over a specified time interval is measured at the following time points: before the start of cooling, 5 minutes into cooling, 15 minutes after the start of cooling, and 10 minutes after rewarming. The ultrasound probe is placed 1 centimeter proximal to the styloid process of the right radius, to evaluate changes in blood flow.
  Unit: Centimeters per second (cm/s)
Time-Averaged Mean Velocity (TAMEAN) | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  The average blood flow velocity in the right radial artery over a specified time interval is measured at the following time points: before the start of cooling, 5 minutes into cooling, 15 minutes after the start of cooling, and 10 minutes after rewarming. The ultrasound probe is placed 1 centimeter proximal to the styloid process of the right radius, to assess changes in blood flow.
  Unit: Centimeters per second (cm/s)
Pulsatility Index (PI) | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  A dimensionless index measuring changes in blood flow velocity over the cardiac cycle is measured at the following time points: before the start of cooling, 5 minutes into cooling, 15 minutes after the start of cooling, and 10 minutes after rewarming. The ultrasound probe is placed 1 centimeter proximal to the styloid process of the right radius, to comprehensively assess changes in arterial vascular function and hemodynamics.
Resistance Index (RI) | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  The Resistance Index (RI) is measured at the following specific time points: before the start of cooling therapy, 5 minutes into the cooling therapy, 15 minutes after the start of cooling therapy, and 10 minutes after the rewarming period. This index is used to assess the resistance to blood flow within the artery and to understand changes in the blood flow status.
Systolic/Diastolic Ratio (S/D) | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  The ratio of systolic to diastolic blood flow velocities is calculated at the following time points: before the start of cooling, 5 minutes into cooling, 15 minutes after the start of cooling, and 10 minutes after rewarming, which helps to assess changes in hemodynamics and vascular health.
Blood Flow Volume (VolFlow) | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  The volume of blood flowing through the right radial artery is measured at the following time points: before the start of cooling, 5 minutes into cooling, 15 minutes after the start of cooling, and 10 minutes after rewarming. The ultrasound probe is placed 1 centimeter proximal to the styloid process of the right radius, to evaluate changes in blood flow.
  Unit: Milliliters per minute (mL/min)
Vessel Diameter (Vas Diam) | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  The internal diameter of the right radial artery is measured before the start of cooling therapy, 5 minutes into cooling, 15 minutes after the start of cooling, and 10 minutes after rewarming. The ultrasound probe is placed 1 centimeter proximal to the styloid process of the right radius to assess the width of the artery lumen.
  Unit: Millimeters (mm)
Vessel Area (Vas Area) | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  The cross-sectional area of the right radial artery is measured at the following time points: before the start of cooling, 5 minutes into cooling, 15 minutes after the start of cooling, and 10 minutes after rewarming. The ultrasound probe is placed 1 centimeter proximal to the styloid process of the right radius, providing an indicator of the artery's size.
  Unit: Square millimeters (mm²)
Room Temperature (°C) | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  Measured at the following time points: before initiation of cooling therapy, 5 minutes after cooling therapy initiation, 15 minutes after cooling therapy initiation, and 10 minutes after rewarming. Unit: degrees Celsius (°C).
Skin Temperature at the Right Brachial Plexus Superficial Ice Pack Application Area (°C) | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  Measured at the following time points: before initiation of cooling therapy, 5 minutes after cooling therapy initiation, 15 minutes after cooling therapy initiation, and 10 minutes after rewarming. Unit: degrees Celsius (°C).
Skin Temperature at the Right Radial Artery Puncture Site (°C) | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  Measured at the following time points: before initiation of cooling therapy, 5 minutes after cooling therapy initiation, 15 minutes after cooling therapy initiation, and 10 minutes after rewarming. Unit: degrees Celsius (°C).
Superficial Skin Temperature at the Left Radial Artery (°C) | From 0 to 3 hours after the volunteers enter the pre-anesthesia holding area.
  Measured at the following time points: before initiation of cooling therapy, 5 minutes after cooling therapy initiation, 15 minutes after cooling therapy initiation, and 10 minutes after rewarming. Unit: degrees Celsius (°C).
Complication | From 0 to 24 hours after the volunteers enter the pre-anesthesia holding area.
  Observe whether there is frostbite in the remote local peripheral nerve cooling treatment, test and puncture area, and diagnose and treat frostbite as early as possible.

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, ph.D, Study Chair — The Second Affiliated Hospital, Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email.
Supporting Information: Study Protocol, SAP, ICF, CSR